CLINICAL TRIAL: NCT05419089
Title: The Sinai Robotic Surgery Trial in HPV-related Oropharyngeal Squamous Cell Carcinoma (SIRS 2.0 Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Raymond Chai, Associate Professor of Otolaryngology, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY 22-00279
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: HPV-positive Oropharyngeal Squamous Cell Carcinoma
Keywords: Oropharyngeal squamous cell carcinoma; OPSCC; Human papillomavirus; Transoral robotic surgery; TORS; HPV; p16; ctDNA; circulating tumor DNA; cfHPVDNA
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Intervention Model Description: Non-randomized non-inferiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic surgery only (Experimental): * Complete resection to negative frozen section margins (pT1-2)
  * < 4 nodes, ≤ 2 mm extranodal extension (ENE), no supraclavicular nodes
  Interventions: Procedure: Robotic surgery

INTERVENTIONS:
Procedure: Robotic surgery — Transoral robotic surgical resection of the tumor with negative intraoperative frozen section margins.

SUMMARY:
The purpose of this study is to determine whether treatment of HPV-related oropharyngeal squamous cell carcinoma in patients with undetectable postoperative HPV circulating tumor DNA (cfHPVDNA) with transoral robotic surgery (TORS) alone can result in cancer control and survival comparable to those previously reported with standard therapy. The protocol includes patients with only with low or intermediate pathologic risk factors following surgery with detectable pre-surgery cfHPVDNA and undetectable post-surgery cfHPVDNA.

The hope is that with this approach, the long-term complications from chemotherapy and radiation can be reduced.

DETAILED DESCRIPTION:
There has been significant increase in the incidence of oropharynx cancer in North America and Europe. It is now understood that there are two dominant carcinogenic pathways for oropharyngeal squamous cell carcinoma. Environmentally related which is caused mainly by smoking and alcohol, and HPV-related oropharyngeal squamous cell carcinoma (HPVOPSCC). HPVOPSCC now accounts for over 80% of OPC seen in the USA and an increasing fraction of these malignancies in Europe. It has been shown that HPVOPSCC confers an excellent prognosis for intermediate staged disease and this has called into question the rational for aggressive concurrent chemoradiotherapy. High-dose radiotherapy (RT) and chemoradiotherapy (CRT) have substantial impact on local tissues and organ function and result in a significant rate of late mortality and morbidity. Studies are now being designed to reduce the impact of RT and CRT for patients.

Recently, a new test has been developed that measures HPV circulating tumor DNA (cfHPVDNA) in the blood. The test has emerged as a promising biomarker for HPVOPSCC, correlating with both treatment response as well as surveillance for cancer recurrence. Data suggests that a negative test in the surveillance period following treatment is highly sensitive and specific for recurrent disease.

In this trial, the study will be stratifying p16 positive patients with PCR detectable high-risk (HR) HPV DNA or RNA following TORS into risk groups based on final pathology to determine appropriate treatment intensity. Patients with low- or intermediate-risk pathologic disease and undetectable postoperative cfHPVDNA will receive no adjuvant therapy. This group includes patients with AJCC 7th edition T1-T2N0-2b disease. Patients must have less than four pathologic nodes on final pathology, negative margins, and no contralateral nodes. Perineural or lymphovascular alone is allowed but not in combination. Microscopic extranodal extension (less than or equal to 2 mm) is allowed. Patients cannot be active smokers or have a 20 or greater pack year history of smoking.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed and identified resectable primary OPSCC with positive p16 immunohistochemistry, defined as strong and diffuse nuclear and cytoplasmic staining in > 70% of tumor cells. Immunohistochemistry must be performed or reviewed at the central laboratory. P16 status may be determined prior to consent and must be confirmed by surgical specimen if a biopsy is unavailable. HR-HPV status and postoperative cfHPVDNA testing must be performed and resulted prior to treatment assignment. Tissue from the primary site must be available for biomarker studies after surgery.
* Patients enrolled in the trial must have pre-surgery baseline cfHPVDNA using the NavDX assay (Naveris, Cambridge, MA). Detectable baseline cfHPVDNA copy number is defined as ≥ 10 fragments/mL and is required for inclusion in the trial.
* Undetectable cfHPVDNA after surgery. All patients should have a repeat cfHPVDNA test within 1 to 5 weeks post-operatively and prior to treatment assignment. Undetectable cfHPVDNA is defined as < 5 fragments/mL.
* AJCC 7th edition early and intermediate stage (T1N0-2B, T2N0-2B) (non-matted) disease without evidence of distant metastases or gross extranodal extension.
* Age ≥ 18 years at screening
* No previous surgery, radiation therapy, or chemotherapy for head and neck cancer (other than excision/incisional biopsy of the primary site, excisional/incisional nodal biopsy, or tonsillectomy) is allowed at time of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* No active tobacco use (≥1cigarette or cigarette-equivalent per day within the last 5 years) and no cumulative smoking history of >20 pack years. 1 cigar = 4 cigarette-equivalent exposure
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must have adequate bone marrow, hepatic and renal functions as defined below:

  * Platelet count ≥ 90 x 109/l.
  * Hemoglobin ≥ 10 g/dl (may achieve by transfusion).
  * Renal function: eGFR ≥ 50 ml/min

Exclusion Criteria

* Age < 18 years at screening
* Pregnant or breast-feeding women.
* Previous or current malignancies at other sites, except for adequately treated in situ carcinoma of the cervix, basal or squamous cell carcinoma of the skin, thyroid cancer, prostate cancer treated with surgery/radiotherapy, ductal carcinoma in situ of the breast treated with surgery/radiotherapy, or other cancer curatively treated and with no current evidence of disease for at least 3 years.
* Other serious illnesses or medical conditions including but not limited to:

  * Unstable cardiac disease despite treatment or myocardial infarction within 6 months prior to study entry.
  * History of significant neurologic or psychiatric disorders including severe dementia or poorly controlled seizures
  * Active clinically significant uncontrolled infection
  * Active peptic ulcer disease defined as unhealed or clinically active
  * Active drug addiction including alcohol, cocaine or intravenous drug use defined as occurring within the 6 months preceding diagnosis
  * Severe chronic obstructive pulmonary disease, defined as being associated with a hospitalization for pneumonia within 12 months of diagnosis.
  * Prior organ transplant
  * Interstitial lung disease
  * Concurrent treatment with any other anti-cancer therapy
  * Participation in an investigational therapeutic drug trial within 30 days of study entry. Participation in additional investigational radiation studies will exclude participation in SIRS. Participation in non-therapeutic, non-oncologic investigational studies (i.e. pain control studies, nutritional studies, etc.) will be allowed amongst SIRS participants, provided there is no alteration of treatment planning, oncologic therapy, or surveillance, and additional studies comply with SIRS safety criteria and stopping rules as outlined in the SIRS protocol.
  * Active hepatitis C by history
* Advanced nodal stage (AJCC 7th edition N2C, N3) or surgically unresectable disease or disease that cannot be fully resected, unequivocal radiographic extranodal extension, unequivocal radiographic or clinical supraclavicular or matted metastatic disease, > 3 unequivocally radiographic pathologic cervical nodes.
* Non-HR-HPV subtype on initial biopsy or final pathology.
* 5 or more positive nodes, irrespective of size, on final pathology.
* p16 or HPV negative OPSCC as determined by IHC and PCR or ISH, respectively.
* Undetectable or < 10 fragments/mL baseline cfHPVDNA prior to surgery.
* Autoimmune disease treated with chemotherapy agents or anti TNF agents within the last 2 years.
* Detectable repeat cfHPVDNA 1-5 weeks postoperatively via the NavDX assay, defined as > 5 fragments/mL.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Local and/or regional disease recurrence (LRR) | 2 years
  Local and/or regional disease recurrence (LRR) at 2 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS at 2 years as defined as the proportion of patients without events (recurrence or death) at 2 years
Disease free survival (DFS) | 2 years
  PFS at 2 years as defined as the proportion of patients without events (recurrence or death) at 2 years
Overall Survival (OS) | 2 years
  OS at 2 years is defined as the proportion of patients alive at 2 years
M.D. Anderson Dysphagia Inventory | 2 years
  20 items instrument: a global assessment (a single question), it comprises three subscales: the emotional subscale (8 items), the functional subscale (5 items), and the physical subscale (6 items). The global assessment refers to the individual's swallowing difficulty as it affects one's overall daily routine. The emotional, functional, and physical subscales refer to the individual's affective response to the swallowing disorder, the impact of the disorder on daily activities, and the self-perception of the swallowing difficulties, respectively. Using a five-point scale (1-5), the minimum total score is 20 and the maximum 100. Higher score indicates the least interference with daily life.
Xerostomia Questionnaire (XQ) | 2 years
  Scale range from 1-10 (1 being dry as a desert and 10 is normal). Higher score indicates better health outcomes
European Organization of Research and Treatment Of Cancer (EORTC QLQ-C30) | 2 years
  EORTC QLQ-C30 is a 30-question tool used to assess the overall QoL in cancer participants. It consisted of 15 domains: 1 GHS/QoL scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). Most items are scored 1 ("not at all") to 4 ("very much") except for the items contributing to the GHS/QoL, which are scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that all transformed scores lie between 0 to 100. For the GHS/QoL and 5 functional scales a high score indicates better global health status/functioning and a negative change from baseline indicated less improvement. Scale ranges from 0-100. For the symptom scales, a high score indicates a higher level of symptoms, and a negative change from baseline indicated an improvement in symptoms.
European Organization of Research and Treatment of Head and Neck cancer questionnaire (EORTC QLQ-H&N35) | 2 years
  EORTC QLQ-H&N35 is a 35-question site-specific tool and is used in conjunction with EORTC QLQ-C30 measurement tool. Scale range from 0-100. Higher score indicates poorer health outcomes.
M.D. Anderson Symptom Inventory - Head & Neck (MDASI-HN) | 2 years
  MDASI-HN is a 28 symptom items questionnaire: 13 general cancer-related symptoms, such as pain, fatigue and nausea; 9 HNC-related symptoms, such as problems with mucus in the mouth and difficulty in swallowing or chewing; 6 items to evaluate the effects of symptoms on daily life, including mood and enjoyment of life. Each item is rated on a 11-point scale from 0 (not at all) to 10 (as bad as you can imagine), while the items that assess the interference of symptoms on daily activities are rated from 0 (does not interfere) to 10 (interfered completely). Subscales and full scale range from 0-10. Higher score indicates poorer health outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Chai, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Valley - Mount Sinai Comprehensive Cancer Care, Paramus, New Jersey
  - Mount Sinai Health System, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.